CLINICAL TRIAL: NCT04986891
Title: Chemotherapy Induced Peripheral Neurotoxicity (CIPN): Why Should we Care (CIPN COST) - Pilot Study
Brief Title: Chemotherapy Induced Peripheral Neurotoxicity (CIPN): Why Should we Care
Acronym: CIPN COST
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: CIPN COST
Record Dates: First submitted 2021-07-15; First posted 2021-08-03 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: CIPN
Keywords: chemotherapy; neuropathy; socio-economic indicators; neurotoxicity; CIPN; quality of life
MeSH Terms: conditions — Neurotoxicity Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- subjects before first chemotherapy cycle with no neuropathy: at least 75 consecutive subjects sent for an evaluation before 1st chemotherapy cycle (TNSc score equal to 0 which means no neuropathy);
- subjects with stable CIPN condition after chemotherapy completion: subjects sent for an evaluation due to stable CIPN condition (CIPN defined as TNSc > or = 1) after chemotherapy completion (at least 2 months off treatment).

SUMMARY:
This is a pilot, observational, cross-sectional, study on socio-economic burden related to chemotherapy-induced peripheral neurotoxicity (CIPN). Investigators will collect CIPN healthcare related costs on a detailed clinical patient-level. As a sub-study, data obtained in this cross-sectional study, will be compared with administrative larger datasets on patients affected by cancer. The aim is to run a test for potential proxy variables which are available in larger administrative datasets, even if not directly measuring CIPN, to learn more about the impact of CIPN.

DETAILED DESCRIPTION:
This is an observational, cross-sectional, pilot study of chemotherapy-induced peripheral neurotoxicity (CIPN) patients, aiming at ascertaining the socio-economic burden related to CIPN.

The study will collect the following information:

* General medical and oncological history
* Neurological assessment formalized via:

  * NCI-CTC v.5 sensory and motor
  * PI-NRS
  * DN4
  * TNSc©
  * Jamar grooved Pegboard test
* Patient reported outcome measures related to CIPN:

  * FACT-GOG NTX v.4©
  * EORTC CIPN20©
* Socio-economic framework: demographic characteristics and working conditions

A sub-study is also planned. For this purpose, a comparison with administrative databases, and in particular the data related to cancer patients, will be performed. Unlike the data adopted in the main analysis of the cross-sectional study, the data provided by administrative datasets do not include direct information on CIPN. Investigators will study whether administrative datasets include variables that could be adopted as proxy for CIPN. It will test the reliability of these proxy variables by comparing the expected distribution of CIPN patients in the latter dataset, with the observed distribution in the outpatient dataset - given specific characteristics of the patients. An analysis of this kind would support the activity of policy makers engaged in the treatment of cancer-related problems.

Study Design: at least 75 consecutive patients who suffer from CIPN and at least 75 consecutive patients before chemotherapy will be enrolled to gain precise information on CIPN severity and its impact on socio-economic indicators. Subjects will be evaluated once, after obtaining written informed consent. A trained investigator will perform the selected healthcare-assessed scales and supervise the patient-completed measures.

ELIGIBILITY:
Inclusion Criteria:

1. Cancer patients with this characteristics:

   1. at least 75 consecutive subjects sent for a neurological evaluation before 1st chemotherapy cycle (TNSc score equal to 0 which means no neuropathy);
   2. at least 75 consecutive subjects sent for a neurological evaluation due to stable CIPN condition (CIPN defined as TNSc > or = 1) after chemotherapy completion (at least 2 months off treatment).
2. Male and female subjects who are 18 years of age or older.
3. Subjects freely provide informed consent by signing and dating an informed consent form prior to study entry.
4. Subjects must be willing to complete all study-related activities and follow-up visits required by the protocol.
5. Subjects must have a Karnofsky performance score greater than or equal to 70.

Exclusion Criteria:

1. Concomitant neurologic conditions (e.g., brain tumor, spinal or brain metastases) that would interfere or complicate the assessments.
2. Severe depression that in the opinion of the Investigator would complicate the assessments.
3. Subjects who are currently receiving another medication other than antineoplastic chemotherapy drugs that has known potential to produce neurologic peripheral nerve toxicity (e.g., metronidazole, isoniazid, amiodarone, antiretroviral medications).
4. Subjects who suffer from another medical condition that can cause neuropathy (e.g., diabetes)
5. Subjects with any other condition, which, in the investigator's judgment, might decrease the chance of obtaining satisfactory data to achieve the objectives of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients (at least 18 years old) as follows. Group A: at least 75 consecutive subjects sent for an evaluation before 1st chemotherapy cycle (TNSc score equal to 0 which means no neuropathy); Group B: at least 75 consecutive subjects sent for an evaluation due to stable CIPN condition (CIPN defined as TNSc > or = 1) after chemotherapy completion (at least 2 months off treatment).
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-07-31 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Correlation between Chemotherapy-induced peripheral neurotoxicity (CIPN) as assessed by Total Neuropathy Score (TNSn©) scale and demographic and socio-economic indicators | Baseline
  Correlation between CIPN (as assessed by TNSn© scale) and demographic and socio-economic indicators collected with a questionnaire filled in at screening. The questions included in the questionnaire are drawn from the national sample surveys by the Ministry of Labor and Social Policies (INAPP) and by the Bank of Italy (SHIW).

SECONDARY OUTCOMES:
Correlation between CIPN as assessed by National Cancer Institute-Common Toxicity Criteria (NCI-CTC v. 5) sensory and motor grade and demographic and socio-economic indicators | Baseline
  Correlation between CIPN assessed by NCI-CTC v.5 sensory and motor questionnaire (0-5 score. where 5 means worse outcome) and demographic and socio-economic indicators collected with a questionnaire filled in at screening.
Correlation between CIPN as assessed by Pain Intensity Numerical Rating Scale (PI-NRS) and demographic and socio-economic indicators | Baseline
  Correlation between CIPN assessed by PI-NRS scale (0-10 score, where 10 means worse outcome) and demographic and socio-economic indicators collected with a questionnaire filled in at screening.
Correlation between CIPN as assessed by Douleur Neuropathique 4 (DN4) scale and demographic and socio-economic indicators | Baseline
  Correlation between CIPN assessed by DN4 scale (0-10 score, where 10 means worse outcome) and demographic and socio-economic indicators collected with a questionnaire filled in at screening.
Correlation between CIPN as assessed by Functional Assessment of Cancer Therapy/Gynecologic Oncology Group - Neurotoxicity 4 (FACT-GOG NTX v.4©) scale and demographic and socio-economic indicators | Baseline
  Correlation between CIPN assessed by FACT-GOG NTX v.4© scale (0-44 score, where 44 means worse outcome) and demographic and socio-economic indicators collected with a questionnaire filled in at screening.
Correlation between CIPN as assessed by European Organization for Research and Treatment of Cancer (EORTC) CIPN20© scale and demographic and socio-economic indicators | Baseline
  Correlation between CIPN assessed by EORTC CIPN20© scale (0-100 score, where 100 means worse outcome) and demographic and socio-economic indicators collected with a questionnaire filled in at screening.
Correlation between CIPN as assessed by Jamar grooved Pegboard test and demographic and socio-economic indicators | Baseline
  Correlation between CIPN assessed by Jamar grooved Pegboard test and demographic and socio-economic indicators collected with a questionnaire filled in at screening.

OTHER OUTCOMES:
To investigate whether the larger administrative datasets include variables that could be adopted as proxy for CIPN | Entire study duration (approximately 8 months)
  Reliability of these proxy variables will be tested by comparing the expected distribution of CIPN patients, in the administrative datasets, with the observed distribution in the cross-sectional study.

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Monza, Monza, Italy

IPD SHARING:
Plan to Share IPD: Undecided